CLINICAL TRIAL: NCT01607684
Title: Pilot Study to Evaluate Magnetic Marker Imaging on Diabetic Polyneuropathy and Gastroparesis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Thomas Seufferlein, Prof. Dr. med., Martin-Luther-Universität Halle-Wittenberg
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PAREMAG; CIV-11-05-000321 (Other: European Databank on Medical Devices - EUDAMED)
Record Dates: First submitted 2012-05-20; First posted 2012-05-30 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-09

CONDITIONS: Diabetic Polyneuropathy; Diabetic Gastroparesis; Diabetes Mellitus
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diabetes mellitus group (Other): Subjects with Diabetes mellitus and symptoms of diabetic gastroparesis
  Interventions: Device: Magnetic Marker Imaging (MMI) with Magma 3D system
- Control group (Other): Healthy volunteers as matched pairs according to gender and age
  Interventions: Device: Magnetic Marker Imaging (MMI) with Magma 3D system

INTERVENTIONS:
Device: Magnetic Marker Imaging (MMI) with Magma 3D system — Magnetic Marker Imaging (MMI). It comprises of a high-resolution three-dimensional detector system, that detects passively and continuously the magnetic field of a magnetic marker capsule (1g, 6x12mm), which is taken orally by the subject. Changes in frequency, intensity and duration of oscillating marker movements allow us to delineate migrating gastric motor complexes. The Magnetic Marker Imaging takes up to 4 h in which the patient lies in a bed. Short interruptions (e.g. to visit the restroom) during this 4 h period are possible.

SUMMARY:
The purpose of this study is to determine whether Magnetic Marker Monitoring is an appropriate opportunity to diagnose and to quantify a suspicious gastroparesis in subjects with diabetic polyneuropathy.

ELIGIBILITY:
Inclusion Criteria:

* age > 50 years
* written informed consent
* Diabetes mellitus (only Diabetes mellitus group)
* Symptoms of diabetic gastroparesis with respect to nausea, postprandial fullness, abdominal pain, nausea, vomiting, abdominal bloating, early satiety, erratic blood glucose levels and weight loss evaluated by a standardized questionnaire (only Diabetes mellitus group)
* actually measured HbA1c (only Diabetes mellitus group)

Exclusion Criteria:

* Subject who is pregnant or breast feeding.
* Subject unwilling or unable to comply with study requirements.
* Any investigational agent or participation in another clinical trial within 28 days prior to randomization
* Any kind of disorder that compromises the ability of the subject to give written informed consent and/or comply with the study procedures.
* History of any medical condition that may increase the risks associated with study participation or may interfere with the interpretation of the study results.
* Known allergy to the investigational product, to any of its excipients
* Active inflammatory bowel disease, serious gastric ulceration or other bowel diseases like e.g. coeliac disease
* Implanted cardiac cardioverter-defibrillator or cardiac pacemaker
* Stenosis or stricture of gastrointestinal tract or any surgery in this region except for cholecystectomy or appendectomy
* Long-term medication with drug, that influence gastrointestinal motility (opiate, opioids, erythromycin, metoclopramide, laxatives) < 3 days before randomisation and before magnetic marker monitoring

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Frequency of gastric peristalsis | 4 hours

SECONDARY OUTCOMES:
Intensity of gastric peristaltic waves | 4 hours
Correlation with other parameters of diabetic polyneuropathy (nausea, postprandial fullness, abdominal pain, nausea, vomiting, abdominal bloating, early satiety, erratic blood glucose levels and weight loss evaluated by a standardized questionnaire) | 4 hours
Influence of age on parameters of diabetic polyneuropathy measurable by magnetic marker imaging | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Seufferlein, MD, Principal Investigator — Martin-Luther-Universität Halle-Wittenberg
Locations (1):
- Universitätsklinikum Halle, Halle, Germany